CLINICAL TRIAL: NCT02061839
Title: Prevention of Melasma Relapse During Summertime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Pharmacologie Clinique Applique a la Dermatologie (Other)
Collaborators: BIODERMA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013-A00073-42
Record Dates: First submitted 2014-02-10; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teinted sunscream (Experimental): UVA, UVB and visible light protection (exactly the same UVA and UVB protection as the comparator)
  Interventions: Other: Sunscream with visible light protection
- Regular sunscream (Active Comparator): UVA and UVB protection
  Interventions: Other: Sunscream

INTERVENTIONS:
Other: Sunscream with visible light protection
  Arms: Teinted sunscream
Other: Sunscream
  Arms: Regular sunscream

SUMMARY:
Main objective is to show that a photoprotective sunscreen having a protection against the visible light is more effective than a sunscreen having the same UVA AND UVB protection but with a low (weak) protection against the visible, to prevent the relapses of the melasma during the summertime.

DETAILED DESCRIPTION:
40 melasma affected women will be included and randomized in two parallel groups (one group protected by a UVA+UVB+visible extended sunscreen and one group group protected by a UVA+UVB sunscreen).

There will be 3 visits: Baseline, T2.5months and T5months (final visit).

Products application frequency: twice daily(morning and afternoon) and additional applications every 2 hours in case of solar exposure.

Main evaluation criterion: the MASI score assessed from standardized photographs (system VISIA, Canfield Scientific, USA) at Baseline, middle and end of study.

ELIGIBILITY:
Inclusion Criteria:

* Melasma

Exclusion Criteria:

* Other pigmentary disorders associated (including PIH)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Comparison between MASI scores before prevention treatment and after 6 months | 6 months
  MASI scores are evaluated by two physicians blinded to the treatment received on standardized pictures taken before treatment and after 6 months of summer period